CLINICAL TRIAL: NCT05075538
Title: COVID-19: Immune Response in Patients With Cancer Undergoing mRNA Vaccination Against SARS-CoV-2
Acronym: I-SPARC
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The population as defined by the inclusion/exclusion criteria and the study logistics were leading to a poor recruitment over the past years.
Sponsor: Jules Bordet Institute (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IJB-COVID-001; 2021-003710-39 (EudraCT Number)
Record Dates: First submitted 2021-10-07; First posted 2021-10-12 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2023-02

CONDITIONS: Cancer
Keywords: immunity; mRNA; vaccination; SARS-CoV-2; COVID-19; COVID19; Spikevax; Comirnaty; Omicron
MeSH Terms: conditions — Neoplasms; COVID-19 | interventions — 2019-nCoV Vaccine mRNA-1273; BNT162 Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Biological: Spikevax — Booster dose, if a booster dose is administered during the study per local / national health policy guidelines.
Biological: Comirnaty — Booster dose, if a booster dose is administered during the study per local / national health policy guidelines.
Biological: Spikevax bivalent Original/Omicron BA.1 — Booster dose, if a booster dose is administered during the study per local / national health policy guidelines.
Biological: Spikevax bivalent Original/Omicron BA.4-5 — Booster dose, if a booster dose is administered during the study per local / national health policy guidelines.
Biological: Comirnaty Original/Omicron BA.1 — Booster dose, if a booster dose is administered during the study per local / national health policy guidelines.
Biological: Comirnaty Original/Omicron BA.4-5 — Booster dose, if a booster dose is administered during the study per local / national health policy guidelines.
Biological: Comirnaty Omicron XBB.1.5 — Booster dose, if a booster dose is administered during the study per local / national health policy guidelines.
Biological: Spikevax Omicron XBB.1.5 — Booster dose, if a booster dose is administered during the study per local / national health policy guidelines.

SUMMARY:
This trial aims to measure the humoral and adaptive immune response in patients with cancer diagnosis undergoing mRNA vaccination against SARS-CoV-2 and assess its efficacy in preventing COVID-19.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old
2. ECOG performance status ≤ 2
3. Subjects with histologically or cytologically confirmed cancer diagnosis (invasive solid tumour or haematological malignancy)

   * undergoing active systemic cancer treatment at the time of the last dose (before ICF signature) of the anti-SARS-CoV-2 mRNA vaccine (such as chemotherapy, immunotherapy, targeted agents, endocrine therapy) in non-metastatic/curative setting or in metastatic/palliative setting
   * or undergoing follow-up after confirmed cancer complete remission without active cancer treatment for the last 12 months at the time of the last dose (before ICF signature ) of the anti-SARS-CoV-2 mRNA vaccine.
4. Life expectancy > 6 months
5. Subjects who received at least 2 doses of mRNA platform vaccination against SARS-CoV-2 as per local guidelines, with the last dose being given between 3 and 12 months prior to baseline assessment.
6. Urine/serum pregnancy test negative for all female subjects of childbearing potential within 7 days prior to subject enrolment.
7. Signed Informed Consent form (ICF) obtained prior to any study related procedure
8. Subject is willing and able to comply with the protocol for the duration of the study including treatment and scheduled visits and examinations.

Exclusion Criteria:

1. Known pregnant and/or lactating women.
2. Subject with a significant medical, neuro-psychiatric, or surgical condition, currently uncontrolled by treatment, which, in the principal investigator's opinion, may interfere with completion of the study.
3. Subjects with active diagnosis of acute leukaemia.
4. Subjects treated with bone marrow transplant < 90 days before received vaccination against SARS-CoV-2.
5. Subjects with a known history of HIV infection.
6. COVID-19 infection in the last 28 days prior to subject enrolment.
7. Subjects receiving prolonged and/or high doses of systemic immunosuppressive therapies including corticosteroids during the last 28 days before receiving first dose of vaccination against SARS-CoV-2 and up to subject enrolment.
8. Subjects who, for any reason, did not receive the 2nd dose of the anti-SARS-CoV-2 mRNA vaccine.
9. Subjects that received the 3rd dose of anti-SARS-CoV-2 mRNA vaccine prior to study entry. Exclusion criterion number 9 is only applicable for previous versions of the protocol and is not applicable from protocol version 3.0 and subsequent versions.
10. Subject that received any dose of non-mRNA anti-SARS-CoV-2 vaccine platform.
11. Subject with a known or suspected history of severe adverse reactions associated with a vaccine and/or with severe allergic reaction to vaccine components or anaphylaxis in the past.
12. Subjects who planned to receive any other licensed vaccines for other indications within 28 days prior to the first booster dose after ICF signature or who are planning to receive any other vaccine up to 14 days after the first booster dose of the mRNA anti-SARS-CoV-2 vaccine after ICF signature (28 days for live attenuated vaccines). For influenza vaccination, a shorter interval or simultaneous administration is acceptable.
13. Subjects who have planned to receive a booster dose after ICF signature but before the baseline assessment
14. Subjects who received COVID-19 pre-exposure prophylactic monoclonal antibodies or who have been treated with anti-SARS-CoV-2 monoclonal antibodies or COVID-19 convalescent plasma during the last 6 months before ICF signature.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2024-01-08 (Actual); Study Completion 2024-01-08 (Actual)

PRIMARY OUTCOMES:
Humoral immune response against SARS-CoV-2 after the last dose of a mRNA anti-SARS-CoV-2 vaccine (Baseline assessment) | 3 to 12 months after the last dose
  Rate of humoral immune response against SARS-CoV-2 between 3 and 12 months after the last dose (before ICF signature) of a mRNA anti-SARS-CoV-2 vaccine (baseline assessment)

SECONDARY OUTCOMES:
Humoral immune response against SARS-COV-2 | at 6 months (+/- 4 weeks) after the baseline assessment or at 6 months (+ 4 weeks/- 8 weeks) after the first booster after ICF signature, if a booster dose of the vaccine is administered during the study per local / national health policy guidelines.
  Duration of humoral immune response against SARS-COV-2 based on the final study assessment, namely at 6 months (+ /- 4 weeks) after the baseline assessment or at 6 months (+ 4 weeks/- 8 weeks) after the first booster dose after ICF signature, if a booster dose of the vaccine is administered during the study per local / national health policy guidelines.
Humoral immune response against SARS-COV-2 by cohort | 3 to 12 months after the last dose before ICF signature; and 6 months (+/- 4 wks) after baseline assessment or 6 months (+ 4 wks/-8 wks) after the first booster after ICF signature if a booster dose is administered during the study
  Rate of humoral immune response against SARS-COV-2 by cohort
Rate of asymptomatic subjects with SARS-CoV-2 positive test during the study | Retrospectively collected at each visit: at baseline assessment, pre-boosting (within 2 wks before 1st booster dose after ICF signature), post-boosting (2 wks after this booster); and 6 months after this booster OR after baseline assessment if no booster
  Rate of asymptomatic subjects with SARS-CoV-2 positive test, confirmed COVID-19 or severe COVID-19 infection with onset at least 14 days after the last dose before ICF signature in subjects who had been without serologic or virological evidence of SARS-CoV-2 infection up to 14 days after the last dose before ICF signature.
Safety of booster dose(s) of mRNA anti-SARS-CoV-2 vaccine received after ICF signature | During the 30 days following the administration of the booster received during the study period (if any)
  Frequency, duration and severity of adverse reactions reported according to NCI Common Terminology Criteria for Adverse Events signature (CTCAE) Version 5.0, if booster dose(s) of the vaccine are administered during the study per local / national health policy guidelines.

OTHER OUTCOMES:
Rate of humoral immune response against SARS-COV-2 before and after the last dose | within 2 weeks before the first booster after ICF signature, at 2 weeks +/- 3 days after the first booster after ICF signature) if a booster dose is administered during the study per local/national health policy guidelines
  Rate of humoral immune response against SARS-COV-2 at pre- (within 2 weeks before the first booster after ICF signature) and post-boosting (at 2 weeks +/- 3 days after the first booster after ICF signature) if a booster dose is administered during the study per local/national health policy guidelines.
Changes in the levels of circulating cytokines/chemokines and the balance or differentiation/activation status of lymphocyte subpopulations and their association with anti-SARS-CoV-2 antibodies | i) 3 to 12 months after the last dose before ICF signature; AND ii) in case of booster before ICF signature, 2 wks before the first booster, 2 wks after this booster, 6 months after this booster OR iii) if no booster 6 months after baseline assessment
  Changes in the levels of circulating cytokines/chemokines and the balance or differentiation/activation status of lymphocyte subpopulations and their association with anti-SARS-CoV-2 antibodies

CONTACTS AND LOCATIONS:
Locations (2):
- Belgium (2):
  - Institut Jules Bordet, Anderlecht
  - CHU UCL Namur Sainte-Elisabeth, Namur